CLINICAL TRIAL: NCT05471661
Title: Administration of Rapidly Generated Multipathogen-specific T-Lymphocytes for the Treatment of AdV, CMV, EBV, BKV and Aspergillus Fumigatus Infections Post Allogeneic Stem Cell Transplant
Brief Title: T Lymphocytes for the Treatment of AdV, CMV, EBV, BKV and Aspergillus Fumigatus Infections After Allogeneic Stem Cell Transplantation
Acronym: Penta-STs-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: George Papanicolaou Hospital (Other)
Collaborators: University General Hospital of Patras (Other)
Responsible Party: Principal Investigator, Evangelia Yannaki, PI, Director of the Gene and Cell Therapy Center, Hematology-HCT Unit, George Papanicolaou Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Penta-STs-001
Record Dates: First submitted 2022-07-16; First posted 2022-07-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Opportunistic Fungal Infection; Opportunistic Viral Infection; Bone Marrow Transplant Infection
Keywords: CMV; EBV; BK virus; Adenovirus; Aspergillus Fumigatus
MeSH Terms: conditions — Adenoviridae Infections

STUDY DESIGN:
Intervention Model Description: Patients from Hematology Department- Hematopoietic Stem Cell Transplantation Unit, George Papanikolaou Hospital and Bone Marrow Transplantation Unit of the University Hospital of Patras will be eligible to receive penta-STs as treatment for infection of one or more of the target-pathogens or for increasing pathogen load in two consecutive timepoints, following any type of allogeneic transplant.
  If patients are receiving steroids for treatment of GVHD or for other reasons, dosage must have been tapered to ≤0.5mg/kg prednisone (or equivalent) prior to study enrollment. Patients may not have received ATG, or Campath or other immunosuppressive monoclonal antibodies in the last 28 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Penta-STs (Experimental): Patients will receive penta-STs in a single infusion. If they have a partial response or receive therapy post-infusion which could ablate the infused T cells they are eligible to receive up to 2 additional doses from 28 days after their first dose.
  Interventions: Biological: Pentavalent-specific T cells (penta-STs)

INTERVENTIONS:
Biological: Pentavalent-specific T cells (penta-STs) — Patients will receive penta-STs in a single infusion. If they have a partial response or receive therapy post-infusion which could ablate the infused T cells they are eligible to receive up to 2 additional doses from 28 days after their first dose.

SUMMARY:
The purpose of the study is to determine the feasibility, safety and efficacy of administering rapidly-generated donor-derived pentavalent-specific T cells (Penta-STs) to mediate antiviral and antifungal activity in hematopoietic stem cell transplant (HSCT) recipients with AdV, EBV, CMV, BKV or Aspergillus fumigatus (AF) infection/ reactivation or with active disease.

DETAILED DESCRIPTION:
Reconstitution of anti-viral and antifungal immunity by donor-derived antigen-specific T cells has shown promise in preventing and treating infections with CMV, or/and EBV, or/and AdV or/and BKV, HHV6 or/and AF post-transplant. However, the broader implementation of T cell immunotherapy using conventional protocols is limited and until today it was practically impossible for Greece by the cost, the complexity and the time required for virus-specific T cells (VSTs) production and by the antigenic competition between different antigens, which limits the spectrum of viruses that can be targeted in a single T cell product.

In this trial, the investigators will evaluate the feasibility, safety and efficacy of donor-derived Penta-STs infusion to allogeneic HSCT recipients with confirmed AdV, EBV, CMV, BKV and AF infection.

ELIGIBILITY:
Inclusion Criteria:

1. Received prior myeoloablative or nonmyeloablative allogeneic hematopoietic stem cell transplant.
2. Cells administered as treatment for single or multiple infections/reactivations of one or more of the following pathogens: AdV, CMV, EBV, ΒΚV and AF.
3. Karnofsky/Lansky score of ≥ 50.
4. ANC > 500/μl.
5. Bilirubin ≤ 2x*, AST < 3x*, Serum creatinine ≤ 2x*, Hemoglobin > 8.0 g/dl.
6. Pulse oximetry of > 90% on room air.
7. Available pentavalent-specific T cells.
8. Negative pregnancy test (if female of childbearing potential)
9. Patient capable of providing informed consent.

Exclusion Criteria:

1. Received ATG, or Campath or other T cell immunosuppressive monoclonal antibodies in the last 28 days.
2. Steroids > 0.5 mg/kg/day prednisone.
3. Received donor lymphocyte infusion in last 28 days.
4. GVHD ≥ grade 2.
5. Active and uncontrolled relapse of malignancy.
6. Patients with other uncontrolled infections

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Acute GvHD | Within 6 weeks post the last dose of penta-STs
  The safety of cell therapy with penta-STs will be assessed according to acute and chronic GvHD grades III-IV
Chronic GvHD | Within 6 months post the last dose of penta-STs
  The safety of cell therapy with penta-STs will be assessed according to acute and chronic GvHD grades III-IV
Infusion-related adverse events | Within 30 days of the last dose of penta-STs
  The safety of cell therapy with penta-STs will be assessed according to grades ≥3 infusion-related adverse events
Non hematological, adverse events | Within 30 days of the last dose of penta-STs
  The safety of cell therapy with penta-STs will be assessed according to grades ≥3 non hematological, adverse events within 30 days of the last penta-ST dose, which are not due to the preexisting infection/comorbidities or the original malignancy
Resolution of infection - 1 | 12 weeks post the last dose of penta-STs
  The efficacy of penta-STs will be determined based on the reduction/elimination of pathogen load in patients with infections
Resolution of infection - 2 | 12 weeks post the last dose of penta-STs
  The efficacy of penta-STs will be determined based on the amelioration/elimination of clinical symptoms in patients with viral disease
Antiviral immunity | 12 weeks post the last dose of penta-STs
  The efficacy of penta-STs will be determined based on the reconstitution of antiviral immunity (determination of virus-specific T cells)
Antifungal immunity | 12 weeks post the last dose of penta-STs
  The efficacy of penta-STs will be determined based on reconstitution of antifungal immunity (determination of Aspergillus fumigatus-specific T cells)
Viral reactivations or recurrence of AF infection | 6 months post the last dose of penta-STs
  The efficacy of penta-STs will be determined by the absence of viral reactivations or recurrence of AF infection post penta-STs infusion

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Yannaki, MD, Principal Investigator — George Papanicolaou Hospital
Locations (2):
- Greece (2):
  - University General Hospital of Patras, Pátrai
  - George Papanikolaou Hospital - Gene and Cell Therapy Center- Hematology Dpt- Hematopoietic Stem Cell Transplant Center, Thessaloniki

IPD SHARING:
Plan to Share IPD: No